CLINICAL TRIAL: NCT03942549
Title: Changes in the Bladder Micro-environment Following Midurethral Sling Surgery for Stress Urinary Incontinence
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: Collins Medical Trust (Other)
Responsible Party: Principal Investigator, Ian Fields, Principal Investigator, Oregon Health and Science University
Other Study IDs: STUDY00019197
Record Dates: First submitted 2019-05-03; First posted 2019-05-08 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Stress Urinary Incontinence
Keywords: microbiome; cytokine
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MUS Cohort: This cohort will undergo midurethral sling placement.
  Interventions: Device: Retropubic midurethral sling

INTERVENTIONS:
Device: Retropubic midurethral sling — Midurethral sling
  Other Names: TVT

SUMMARY:
This observational cohort study is aimed at determining changes in the cytokine expression profile as well as the urinary and vaginal microbiome of women undergoing midurethral sling placement for the treatment of stress urinary incontinence.

DETAILED DESCRIPTION:
Primary Objectives:

This is a pilot study to evaluate how midurethral sling (MUS) placement for the treatment of stress urinary incontinence (SUI) affects the bladder microenvironment, specifically the local microbial community or "microbiome" of the bladder and the cytokine expression profile. The investigators also aim to correlate any changes in the microbiome or cytokine expression profile with patient-reported urinary symptoms preoperatively and postoperatively.

Specific Aim 1: Assess the change in the urinary and vaginal microbiome (preoperatively to postoperatively) in women undergoing MUS placement for the treatment of SUI. The investigators hypothesize that the bladder environment will be disturbed by surgery involving the lower urinary tract and will show demonstrable changes in the urinary and vaginal microbiota.

Specific Aim 2: Characterize the cytokine profile of the bladder (preoperatively to postoperatively) in women undergoing MUS placement for the treatment of SUI. The investigators hypothesize that MUS treatment will change the cytokine profile of the bladder and lead to alterations in the expression of pro-inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Planning to undergo retropubic midurethral sling placement

Exclusion Criteria:

* Prior surgery for stress urinary incontinence
* Untreated pelvic organ prolapse > Stage II based on POP-Q assessment
* Concomitant surgery for prolapse
* Current use of anticholinergic medications
* Use of systemic or vaginal antibiotics in the last 2 months
* Active urinary tract infection
* History of recurrent UTI
* Pregnancy
* History of pelvic radiation or bladder cancer

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include women over the age of 18 planning to undergo stand-alone midurethral sling placement for treatment of stress urinary incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Urinary Microbiome | Six weeks
  change in the relative abundance of urinary lactobacillus between baseline, 2 and 6 weeks postoperative

SECONDARY OUTCOMES:
Prevalence of overactive bladder symptoms | Six weeks
  Validated symptom questionnaires will be collected at baseline and again at 2 and six weeks postoperatively to assess common symptoms associated with overactive bladder.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Legacy Good Samaritan Hospital, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No